CLINICAL TRIAL: NCT05765968
Title: Cumulative Live Birth Rates in the Same Cycle Double Stimulation Protocol Versus a Two-cycle Antagonist Stimulation Protocol in IVF Patients With a Poor Prognosis: a Randomized Clinical Trial
Brief Title: Cumulative Live Birth After Double Stimulation Protocol Versus Antagonist Protocol for Poor Ovarian Responders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Hunan Provincial Maternal and Child Health Care Hospital (Other); Jinghua Hospital of Shenyang (Unknown); Xinjiang Jiayin Hospital (Unknown); The Affiliated Hospital of Inner Mongolia Medical University (Other); Guangdong Second Provincial General Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Wuhan Tongji Reproductive Medicine Hospital (Unknown); Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Principal Investigator, Chen Zi-Jiang, Academician, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DouAnt
Record Dates: First submitted 2023-02-28; First posted 2023-03-13 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Infertility
Keywords: Poseidon criteria; Double stimulation; Cummulative live birth
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double Stimulation Protocol (Experimental): Double stimulations were performed during the follicular and luteal phases in the same cycle by rFSH&hmg.
  Interventions: Procedure: Double Stimulation Protocol
- Antagonist Stimulation Protocol (Active Comparator): The classical antagonist protocol were performed by rFSH,hmg and antagonist.
  Interventions: Procedure: Antagonist Stimulation Protocol

INTERVENTIONS:
Procedure: Double Stimulation Protocol — cummulative live birth outcome after two cycles of in virto fertilization using double stimulation protocol, which refers to two cycles of ovarian stimulation in both follicular phase and luteal phase within the same menstrual cycle
  Arms: Double Stimulation Protocol
Procedure: Antagonist Stimulation Protocol — cummulative live birth outcome within no more than two cycles of in virto fertilization using classical antagonist protocol
  Arms: Antagonist Stimulation Protocol

SUMMARY:
To compare the difference in cumulative live birth rates within one year between double stimulations protocol and two-cycle antagonist protocol in poor ovarian responders.

DETAILED DESCRIPTION:
The theory of multicyclic development of follicles during the menstrual cycle prompted new approaches to ovarian stimulation such as double stimulation within the same menstrual cycle, in both follicular and luteal phases. The double ovarian stimulation protocol has been proposed to optimize the number of oocytes retrieved within the shortest possible timeframe.In general, the aim of DUOSTIM is to obtain the highest number of oocytes in the shortest time, thus avoiding waste of time, which is crucial for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Women diagnosed with Poseidon criteria or expected poor ovarian responder （the number of oocyte retrieval ≤9）
2. Women aged ≥20 years old
3. Women who are undergoing their first or second ART cycles
4. Women who are undergoing IVF,ICSI or PGT-A cycles
5. Women with the number of oocyte retrieval ≤9 after their first ovarian stimulation cycle since radomization, and the number of follicle measuring 8mm or larger ≥3

Exclusion Criteria:

1. Women with RIF or RSA
2. Women diagnosed with uterine abnormalities including uterine malformations, adenomyosis, submucosal fibroids, uterine adhesions or endometrial polyps
3. Women with untreated hydrosalpinx that is visible under pelvic ultrasound
4. Women with chromosomal abnormalities, or women who are undergoning PGT-SR or PGT-M cycles
5. Women with a history of canceled FET cycle(s) due to a thin endometrium (<7mm)
6. Man with operation to get sperm

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1198 (Estimated)
Dates: Start 2023-03-14 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative live birth rate | 36 months
  Live birth is defined as the delivery of any viable infant at 28 weeks or more of gestation after our interventions, and cumulative live birth rate is calculated by dividing the number of women achieving live birth after transfers of all study-specific embryos (up to 3 transfers of single blastocycst within 1 year after randomization), by the total number of women randomized to the specific group.

SECONDARY OUTCOMES:
Number of retrieved oocytes | 24 months

OTHER OUTCOMES:
Clinical pregnancy rate | 36 months
  Twenty days after conception, transvaginal ultrasonography will be performed. Clinical pregnancy will be diagnosed with detection of an intrauterine gestational sac.
Incidence of obstetric complications | 36 months
  Number of pregnancies with complications / number of pregnancies.
Incidence of perinatal complications | 36 months
  Number of live births with neonatal complications / number of live births.
Cost-effectiveness analysis | 36 months
  Cost-effectiveness will be evaluated by comparing the two groups in terms of costs and benefits
Birth weight | 36 months
  Weight of newborns at delivery
Total amount of Gn used during ovarian stimulation | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No